CLINICAL TRIAL: NCT07233265
Title: Comparison of Single Incision Scrotal Orchidopexy Versus Standard Two Incision Inguinal Orchidopexy in Children With Palpable Undesended Testis in Children Hospital Faisalabad.
Brief Title: Comparison of Single Incision Scrotal vs Standard Two Incision Inguinal Orchidopexy in Children Under 10 Years.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children Hospital Faisalabad (Other)
Responsible Party: Principal Investigator, Ijaz Ul Haq, Principal investigator, department of paediatric surgery, Children Hospital Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CH-FSD -Orchidopexy- 2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Undescended Testis
Keywords: Orchidopexy; Scrotal incision; Inguinal incision; Paediatric surgery
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single scrotal incision orchidopexy (Experimental): Children in this group undergoes single incision scrotal orchidopexy with palpable undesended testis in superficial inguinal canal.
  Interventions: Procedure: Single scrotal incision orchidopexy
- Standard two incision inguinal orchidopexy (Active Comparator): Children in this group undergoes standard two incision inguinal orchidopexy.
  Interventions: Procedure: Standard two incision inguinal orchidopexy

INTERVENTIONS:
Procedure: Single scrotal incision orchidopexy — Conventional orchidopexy performed through single scrotal incision
  Arms: Single scrotal incision orchidopexy
Procedure: Standard two incision inguinal orchidopexy — Conventional orchidopexy performed through separate inguinal and scrotal incision
  Arms: Standard two incision inguinal orchidopexy

SUMMARY:
This study compares the outcome of single incision scrotal orchidopexy with standard two incision inguinal orchidopexy in children under 10 years of age presented with palpable undesended tesis.The aim is to evaluate operative time,cosmetic outcome and post operative complications.

DETAILED DESCRIPTION:
All patients fulfilling the inclusion criteria admitted to paediatric surgery will be included by after taking informed consent from parents. Patients will be randomized in to two groups by lottery method.In group A ,orchidopexy is performed through single scrotal incision .In group B, orchidopexy is performed through standard two incision inguinal approach. This study compares the outcome interm of operative time, cosmetic outcome and post operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Male children with age 1-10 years. Palpable low -lying undesended tesis.

Exclusion Criteria:

* Impalpable testis Known bleeding disorder

Ages: 12 Months to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Post operative complications | With in 24 hours -1month after surgery .
  Numbers and type of post operative complications (Scrotal hematoma, infection, scrotal edema and testicular atrophy.

SECONDARY OUTCOMES:
Cosmetic outcome | 2 weeks after surgery
  Cosmetic appearance of surgical scar assessed by standardized scale. Scale score range (1-10) lower score =better cosmetic outcome. Higher core = worse cosmetic outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital and Institute of Child Health Faisalabad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No